CLINICAL TRIAL: NCT03436277
Title: Effect of the Administration of L-Carnitine on Body Fat Percentage and Body Weight in Overweight Women in Crossfit Training.
Brief Title: Effect of the Administration of L-Carnitine on Body Weight in Women in Crossfit Training
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Diana Mercedes Hernández Corona, PhD of Pharmacology, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LC-CUT-DMHC
Record Dates: First submitted 2018-02-11; First posted 2018-02-19 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Body Weight Changes
Keywords: Overweight; Obesity; L-Carnitine; Body weight; Body fat percentage
MeSH Terms: conditions — Body Weight Changes; Overweight; Obesity; Body Weight | interventions — Carnitine; trichlorosucrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Sucralose 1,5 g
  Interventions: Dietary Supplement: Sucralose
- L-Carnitine (Experimental): L- Carnitine 1,5 g
  Interventions: Drug: L-Carnitine

INTERVENTIONS:
Drug: L-Carnitine — L-Carnitine oral solution 1.5 g diluted in 250 ml of water, before crossfit training, 5 times a week for 8 weeks
  Other Names: Levocarnitine; Vitamin BT
  Arms: L-Carnitine
Dietary Supplement: Sucralose — Sucralose 1.5 g diluted in 250 ml of water, before crossfit training, 5 times a week for 8 weeks
  Other Names: Trichlorogalacto-sucrose
  Arms: Placebo

SUMMARY:
The L-carnitine has demonstrated effects in the treatment of obesity mainly promoting the fat degradation during exercise.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled clinical trial will be carry out in 24 woman with body mass index ≥ 25 to 29.9 kg/m2. The patients will receive 1.5 g of L-Carnitine deluded in 250 ml of water or placebo before crossfit training, 5 times a week for 8 weeks. Before and after intervention the investigators evaluate: The body composition (body fat, lean body mass), arm muscle circumference, waist circumference, body weight and body mass index.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who practice crossfit regularly (who have 3 months prior to the beginning of the study practicing crossfit).
* Volunteers with a body mass index equal to or greater than 25 Kg/m2.
* Volunteers who do not have allergies to L-Carnitine or any of its components.
* Informed consent signed
* Women with a recommendation of nutrition two weeks prior to the start of the study.
* Body weight stable the last 3 months.

Exclusion Criteria:

* Volunteers with pathologies such as diabetes, hypertension, metabolic syndrome and allergies.
* Women with confirmed or suspected pregnancy.
* Women under lactation and/or puerperium.
* Hypersensibilility to L-Carnitine or Sucralose.
* Kown of renal, hepatic or thyroid deseased.
* Current or previous treatment diet (3 months before inclusion to the study).
* Current pharmacological treatment for loose body weight or 3 months before inclusion to the study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-12-17 (Estimated); Primary Completion 2019-02 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Body Fat | 8 weeks
  Calulated by Durnin formula. Results are reported in percentage and kg
Lean body mass | 8 weeks
  Calulated by Durnin formula. Results are reported in percentage and kg
Body Weight | 8 weeks
  Subject go up onto the scale and stand still over the center of the scale with body weight evenly distributed between both feet. Omron hbf-514c an digital scale and results are reported in kg with a decimal.

SECONDARY OUTCOMES:
Arm muscle circumference | 8 weeks
  The right arm measure to the nearest centimeter with a measuring tape. Then, triceps skinfold thickness, an established measure of fat stores, measure to the nearest millimeter in the right arm using a skinfold caliper
Waist circumference | 8 weeks
  Flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
  Waist circumference was measured with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
  Waist circumference was measured with a flexible tape in the midpoint between the lowest rib and the iliac crest and is expressed in centimeters.
Body Mass Index | 8 weeks
  Body mass divided by the square of the body height, and reported in units of kg/m2.

CONTACTS AND LOCATIONS:
Overall Officials: Diana M Hernández, Principal Investigator — University of Guadalajara
Locations (1):
- Centro Universitario de Tonalá, Tonalá, Jalisco, Mexico

REFERENCES:
- [Background] Huang A, Owen K. Role of supplementary L-carnitine in exercise and exercise recovery. Med Sport Sci. 2012;59:135-142. doi: 10.1159/000341934. Epub 2012 Oct 15. PMID 23075564
- [Background] Villani RG, Gannon J, Self M, Rich PA. L-Carnitine supplementation combined with aerobic training does not promote weight loss in moderately obese women. Int J Sport Nutr Exerc Metab. 2000 Jun;10(2):199-207. doi: 10.1123/ijsnem.10.2.199. PMID 10861338
- [Background] Hongu N, Sachan DS. Carnitine and choline supplementation with exercise alter carnitine profiles, biochemical markers of fat metabolism and serum leptin concentration in healthy women. J Nutr. 2003 Jan;133(1):84-9. doi: 10.1093/jn/133.1.84. PMID 12514272
- [Background] Broad EM, Maughan RJ, Galloway S DR. Effects of exercise intensity and altered substrate availability on cardiovascular and metabolic responses to exercise after oral carnitine supplementation in athletes. Int J Sport Nutr Exerc Metab. 2011 Oct;21(5):385-97. doi: 10.1123/ijsnem.21.5.385. Epub 2011 Aug 3. PMID 21813919
- [Background] Behrend AM, Harding CO, Shoemaker JD, Matern D, Sahn DJ, Elliot DL, Gillingham MB. Substrate oxidation and cardiac performance during exercise in disorders of long chain fatty acid oxidation. Mol Genet Metab. 2012 Jan;105(1):110-5. doi: 10.1016/j.ymgme.2011.09.030. Epub 2011 Oct 1. PMID 22030098
- [Background] Kraemer WJ, Spiering BA, Volek JS, Ratamess NA, Sharman MJ, Rubin MR, French DN, Silvestre R, Hatfield DL, Van Heest JL, Vingren JL, Judelson DA, Deschenes MR, Maresh CM. Androgenic responses to resistance exercise: effects of feeding and L-carnitine. Med Sci Sports Exerc. 2006 Jul;38(7):1288-96. doi: 10.1249/01.mss.0000227314.85728.35. PMID 16826026